CLINICAL TRIAL: NCT04432142
Title: Immune Profiling of Stage III Non-small Cell Lung Cancer Patients Treated With Concurrent Chemoradiation and Adjuvant Durvalumab: A Prospective Observational Phase II Trial
Acronym: IPON-1
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IPON-1
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At five timepoints 60ml of blood will be drawn for biobanking of plasma, serum, and buffy coat samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proton: Patients receiving proton therapy
- Photon: Patients receiving photon therapy in 4 fractions or less

SUMMARY:
Currently, there is only limited data available on the functional immune changes after concurrent chemoradiation in NSCLC (non-small cell lung cancer) patients. Identifying the effect of the treatment on immune cells and what their functional consequences are is an essential first step to come to prognostic and predictive biomarkers.

Many studies investigating the role of immunomodulatory effects of treatment are carried out in either in vitro or in vivo animal models. However, identified factors frequently hamper clinical validation. In addition, as mentioned earlier, although several immunogenic factors have been shown to be released by irradiated tumor cells, so far, only a limited number of studies searched for potential predictive and prognostic immunological biomarkers.

This will be the first time that the immune effects of both treatment modalities will be studied, with, in addition, the immune changes during durvalumab treatment, which are also unknown at present. By getting more insight in the treatment-induced immunomodulatory effects, ultimately, in subsequent projects, this will allow to determine optimal immune stimulation and hence improved outcomes of subsequent durvalumab immune therapy.

DETAILED DESCRIPTION:
Even with the addition of durvalumab to concurrent chemoradiation, approximately only half of the patients are alive at 3 years, and more have progressed already, either locally or distant. Not much is known regarding to identification of patients that will benefit from adjuvant durvalumab, or regarding resistance to adjuvant durvalumab after chemoradiation. Most data on immunotherapy resistance come from metastatic patients treated with monotherapy PD-(L)1 antagonists. Depending on PD-L1 expression level, 10-44% of patients respond well to PD-(L)1 antagonists. The majority of patients are either unresponsive, or experience a tumor recurrence after achieving an initial response. The development of individual immunological treatment strategies (e.g. selection of best treatment: mono- or combination ICI, ICI combined with chemotherapy, or the addition of radiotherapy) is hampered by the lack of knowledge in the best timing, sequencing, and dosing of all modalities and the lack of optimal biomarkers for monitoring the treatment response. This highlights the need of clear biomarkers that can be used to select the best treatment for each individual patient and predict whether patients will benefit from adjuvant immunotherapy. Currently, there is only limited data available on the functional immune changes after concurrent chemoradiation in NSCLC patients. Identifying the effect of the treatment on immune cells (e.g. T-, B-, NK-cells, dendritic cells, macrophages) and what their functional consequences are is an essential first step to come to prognostic and predictive biomarkers.

Many studies investigating the role of immunomodulatory effects of treatment are carried out in either in vitro or in vivo animal models. However, identified factors frequently hamper clinical validation. In addition, as mentioned earlier, although several immunogenic factors have been shown to be released by irradiated tumor cells, so far, only a limited number of studies searched for potential predictive and prognostic immunological biomarkers.

This will be the first time that the immune effects of both treatment modalities will be studied, with, in addition, the immune changes during durvalumab treatment, which are also unknown at present. By getting more insight in the treatment-induced immunomodulatory effects, ultimately, in subsequent projects, this will allow to determine optimal immune stimulation and hence improved outcomes of subsequent durvalumab immune therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of adequately staged (according to standard practice using chest-CT, FDG-PET, brain imaging MRI/CT) NSCLC
* Participant is willing and able to give informed consent for participation in the trial
* Male or female, aged 18 years or above
* Scheduled to receive one of the following two therapeutic strategies:

  * Concurrent chemotherapy and radiotherapy with photons (60 Gy in 30 fractions of 2 Gy) in patients with stage III NSCLC
  * Concurrent chemotherapy and radiotherapy with protons (60 Gy in 30 fractions of 2 Gy) in patients with stage III NSCLC
* Is able and willing to comply with all trial requirement

Exclusion Criteria:

* Mixed non-small cell lung cancer with other histologies such as small cell lung cancer
* Not able to comply with the study protocol
* Less than 18 years' old
* Pregnancy or not able to comply with adequate contraception in women with child baring potential
* Previous radiotherapy to the chest for benign or malignant conditions, including radiation for breast cancer
* Previous malignancy treated with chemotherapy, immune therapy or radiotherapy (irrespective of when this happened)
* Previous malignancies treated with surgery only are allowed if 2 years or more before inclusion in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III NSCLC who are eligible for curative intent concurrent chemotherapy and radiotherapy will be enrolled in the study. They receive standard radiotherapy (60 Gy in 30 fractions of 2 Gy) with protons or photons according to the standard of care. Eligible patients will thereafter receive standard durvalumab immune therapy for 12 months. Eligibility criteria for this study are therefore similar to those for standard of care treatment.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Immune changes | 3 months
  Number of patients with immune changes in stage III NSCLC patients receiving concurrent chemoradiation with protons or photons followed by durvalumab.

SECONDARY OUTCOMES:
PFS | 12 months
  Progression Free Survival
OS | 12 months
  Overall survival
Toxicity chemoradition | until 3 months after chemo/radiotherapy
  - Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 during and after concurrent chemoradiation, also in relation to the irradiated bone marrow volume
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 during courses of Durvalumab | Until 12 months after chemo/radiotherapy
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 of durvalumab and chemoradiation treatment
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Until 12 months after chemoradiation
  Incidence and severity of adverse events (Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 and patient reported outcome (PRO)-CTCAE)
Immune changes compared | Until 12 months after chemoradiation
  Number of patients with immune changes that are distinct for proton therapy compared with photon therapy
Cardiac function | Until 12 months after chemoradiation
  Troponins
Cardiac function | Until 12 months after chemoradiation
  ECG QT Interval
Cardiac function | Until 12 months after chemoradiation
  blood pressure
Cardiac function | Until 12 months after chemoradiation
  BNP
Neurocognitive function test | Until 12 months after chemoradiation
  MOS
Neurocognitive function test | Until 12 months after chemoradiation
  Controlled oral word association
Neurocognitive function test | Until 12 months after chemoradiation
  Trail making test
Neurocognitive function test | Until 12 months after chemoradiation
  HVALT-R test
Tumor material | Until 12 months after chemoradiation
  Obtaining tumor material from standard diagnostic material for translational purposes

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD, PhD, Principal Investigator — Maastro
Locations (1):
- Maastricht Radiation Oncology (MAASTRO clinic), Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No